CLINICAL TRIAL: NCT04015531
Title: Hypofractionated Versus Conventional Fractionation Radiation After Conservative Surgery or Mastectomy With Irradiation of Lymph Node Drainage: a Phase II Randomized Clinical Trial for the Evaluation of Acute Toxicity
Brief Title: Hypofractionated Versus Conventional Fractionation Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital da Baleia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RT 1901
Record Dates: First submitted 2016-08-08; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer; Radiation Toxicity
Keywords: breast cancer; radiotherapy; hypofractionated therapy; nodal irradiation
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Radiation toxicity will be analysed by a blind second investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional radiotherapy (Active Comparator): 50 Gy in 25 fractions to chest wall or whole breast and regional lymph regions (supraclavicular fossa with or without axilla), followed by tumor bed boost of 10 Gy in 5 fractions in case of breast conserving surgery.
  Total time: 5-6 weeks.
  Interventions: Radiation: Conventional radiotherapy
- Hypofractionated radiotherapy (Experimental): 40 Gy in 15 fractions (2.67 Gy each) to chest wall or whole breast and regional lymph regions (supraclavicular fossa with or without axilla).
  Patients undergoing breast conserving surgery will receive concomitant boost with total dose of 48 Gy in 15 fractions (3.20 Gy each) to tumor bed.
  Total time: 3 weeks.
  Interventions: Radiation: Hypofractionated radiotherapy

INTERVENTIONS:
Radiation: Conventional radiotherapy — 50 Gy / 25 fractions / 5-6 weeks / Sequential boost of 10 Gy in 5 fractions, in case of conservative surgery.
  Other Names: Standard fractionation
  Arms: Conventional radiotherapy
Radiation: Hypofractionated radiotherapy — 40 Gy / 15 fractions / 3 weeks / Concomitant boost with total dose of 48 Gy in 15 fractions, in case of conservative surgery.
  Other Names: Hypofractionated therapy
  Arms: Hypofractionated radiotherapy

SUMMARY:
This study was designed to evaluate the acute toxicity and quality of life of hypofractionated radiation versus conventional when regional node irradiation is indicated after breast-conserving surgery or mastectomy.

DETAILED DESCRIPTION:
Investigators hypothesize that hypofractionated radiotherapy is equal effective and safe as conventional radiotherapy in breast cancer patients undergoing regional nodal irradiation.

Eligible breast cancer patients are randomized 1:1 into the following two groups:

1. Hypofractionated therapy: 40 Gy in 15 fractions of 2.67 Gy in breast or chest wall and nodal drainage with Concurrent boost 48.0 Gy / 3.2 Gy daily in tumor bed, in case of conservative surgery;
2. Standard fractionation: 50 Gy in 25 fractions in breast or chest wall and nodal drainage with sequential tumor bed boost with 10 Gy in 5 fractions in tumor bed in case of conservative surgery.

Patients will be followed for 6 months after radiotherapy to evaluate acute toxicity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Older than 18;
* Breast cancer stage T1 - T3;
* At least 1 lymph node positive;
* Treated with mastectomy or conservative surgery;
* Negative surgical margins;
* No distant metastasis;
* No supraclavicular or internal mammary nodes metastases;
* Adjuvant systemic therapy with chemotherapy, endocrine therapy or anti-HER2 (Human - - Epidermal Growth Factor Receptor 2) treatment is accepted;
* Signed informed consent.

Exclusion Criteria:

* Positive surgical margins;
* Concomitant chemotherapy;
* Supraclavicular or internal mammary nodes metastases;
* Distant metastasis;
* Previous thoracic radiotherapy;
* Bilateral breast cancer;
* Patients with collagen diseases;
* Unable or unwilling to sign inform consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
CTCAE Toxicity Assessement - Acute Toxicity | Before treatment, every week of treatment (week 1 to 3 or 1 to 5-6, according to the treatment arm), at the end of treatment (week 3 or week 5-6, according to the treatment arm), 4, 8 and 24 weeks after the last fraction received.
  Change in acute toxicity will be assessed according to criteria of CTCAE version 4.03.

SECONDARY OUTCOMES:
Quality of Life - EORTC QLQ-C30 (version 3) | Before treatment, at the end of treatment (week 3 or week 5-6, according to the treatment arm),1 and 6 months after last fraction received.
  Patients' quality of life will be assessed using self-administered questionnaire EORTC-QLQ-C30 (version 3).
Quality of Life - EORTC breast cancer module (BR23) | Before treatment, at the end of treatment (week 3 or week 5-6, according to the treatment arm),1 and 6 months after last fraction received.
  Patients' quality of life will be assessed using self-administered questionnaire EORTC breast cancer module (BR23).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Oliveira B Gil, MD, Principal Investigator — Baleia Hospital

IPD SHARING:
Plan to Share IPD: Yes
Use of a controlled access approach, with a transparent system to review requests and provide secure data access; assurance that patient privacy and confidentiality can be maintained;
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 2020 onwards
Access Criteria: Principal investigator's e-mail

REFERENCES:
- [Background] Wang SL, Fang H, Song YW, Wang WH, Hu C, Liu YP, Jin J, Liu XF, Yu ZH, Ren H, Li N, Lu NN, Tang Y, Tang Y, Qi SN, Sun GY, Peng R, Li S, Chen B, Yang Y, Li YX. Hypofractionated versus conventional fractionated postmastectomy radiotherapy for patients with high-risk breast cancer: a randomised, non-inferiority, open-label, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):352-360. doi: 10.1016/S1470-2045(18)30813-1. Epub 2019 Jan 30. PMID 30711522
- [Background] EBCTCG (Early Breast Cancer Trialists' Collaborative Group); McGale P, Taylor C, Correa C, Cutter D, Duane F, Ewertz M, Gray R, Mannu G, Peto R, Whelan T, Wang Y, Wang Z, Darby S. Effect of radiotherapy after mastectomy and axillary surgery on 10-year recurrence and 20-year breast cancer mortality: meta-analysis of individual patient data for 8135 women in 22 randomised trials. Lancet. 2014 Jun 21;383(9935):2127-35. doi: 10.1016/S0140-6736(14)60488-8. Epub 2014 Mar 19. PMID 24656685
- [Background] Duxbury PJ, Gandhi A, Kirwan CC, Jain Y, Harvey JR. Current attitudes to breast reconstruction surgery for women at risk of post-mastectomy radiotherapy: A survey of UK breast surgeons. Breast. 2015 Aug;24(4):502-12. doi: 10.1016/j.breast.2015.05.002. Epub 2015 May 26. PMID 26021276
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial A of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet Oncol. 2008 Apr;9(4):331-41. doi: 10.1016/S1470-2045(08)70077-9. Epub 2008 Mar 19. PMID 18356109
- [Background] Shaitelman SF, Schlembach PJ, Arzu I, Ballo M, Bloom ES, Buchholz D, Chronowski GM, Dvorak T, Grade E, Hoffman KE, Kelly P, Ludwig M, Perkins GH, Reed V, Shah S, Stauder MC, Strom EA, Tereffe W, Woodward WA, Ensor J, Baumann D, Thompson AM, Amaya D, Davis T, Guerra W, Hamblin L, Hortobagyi G, Hunt KK, Buchholz TA, Smith BD. Acute and Short-term Toxic Effects of Conventionally Fractionated vs Hypofractionated Whole-Breast Irradiation: A Randomized Clinical Trial. JAMA Oncol. 2015 Oct;1(7):931-41. doi: 10.1001/jamaoncol.2015.2666. PMID 26247543
- [Background] Bekelman JE, Sylwestrzak G, Barron J, Liu J, Epstein AJ, Freedman G, Malin J, Emanuel EJ. Uptake and costs of hypofractionated vs conventional whole breast irradiation after breast conserving surgery in the United States, 2008-2013. JAMA. 2014 Dec 17;312(23):2542-50. doi: 10.1001/jama.2014.16616. PMID 25494006
- [Background] Jagsi R, Falchook AD, Hendrix LH, Curry H, Chen RC. Adoption of hypofractionated radiation therapy for breast cancer after publication of randomized trials. Int J Radiat Oncol Biol Phys. 2014 Dec 1;90(5):1001-9. doi: 10.1016/j.ijrobp.2014.09.032. PMID 25539365